CLINICAL TRIAL: NCT00130000
Title: SHEPHERD: Safety in Hemolytic PNH Patients Treated With Eculizumab: A Multi-Center Open-Label Research Design
Brief Title: Eculizumab to Treat Paroxysmal Nocturnal Hemoglobinuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050217; 05-H-0217
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-06-25

CONDITIONS: Paroxysmal Hemoglobinuria, Nocturnal
Keywords: h5g.1; Paroxysmal Nocturnal Hemoglobinuria; SHEPHERD; PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

INTERVENTIONS:
Drug: Eculizumab

SUMMARY:
This study will evaluate the safety and effectiveness of the experimental drug eculizumab for treating paroxysmal nocturnal hemoglobinuria (PNH), a disorder that can cause premature destruction of red blood cells. PNH may result in anemia requiring blood transfusions. Patients may be at high risk of life-threatening blood clots in their veins and may have urine discoloration, stomach pain, difficulty swallowing, tiredness, and poor quality of life. Men may have problems getting or maintaining an erection. Eculizumab is a monoclonal antibody that may improve the survival of red blood cells in patients with PNH.

Patients 18 years of age and older who have been diagnosed with PNH for more than 6 months, who have active disease, and who require blood transfusions may be eligible for this study. Each candidate is screened with a physical examination, electrocardiogram, blood and urine tests, and a questionnaire for information on how PNH affects the patient physically, socially, emotionally, and functionally.

Participants receive infusions of eculizumab through a needle in a vein once a week for five doses and then every two weeks for another 24 doses. All patients are vaccinated against Neisseria meningitides, a bacteria that can cause symptoms, possibly including life-threatening meningitis, in susceptible people, including people who take eculizumab.

At every treatment visit, patients update their health status, transfusion record, and medication use; review their laboratory results from the preceding visit; have vital signs measured; and provide a blood sample for laboratory tests. At selected visits, they also provide a urine sample, have a repeat electrocardiogram, and complete a questionnaire. At the final treatment visit, participants have a complete physical examination, in addition to the routine procedures.

DETAILED DESCRIPTION:
Paroxysmal nocturnal hemoglobinuria (PNH) is an acquired clonal disorder of the hematopoietic stem cell characterized by intravascular hemolysis, hemoglobinuria, anemia, and thrombosis. The clinical features of PNH result from the lack of one or more of GPI-linked proteins that serve to protect cells from autologous complement mediated attack. Two such proteins, CD55 (decay accelerating factor) and CD59 (reactive lysis inhibitor) have been shown to be absent from PNH erythrocytes and platelets as well as other cell types.

Evidence strongly suggests that lack of the terminal complement inhibitor CD59 is responsible for the sensitivity of PNH erythrocytes and platelets to the effects of autologous complement. Since the pathogenesis of PNH is due to the inability of PNH red cells and platelets to inhibit the activation of terminal complement, it is logical to hypothesize that a terminal complement inhibitor could effectively stop the intravascular hemolysis, obviate or lessen the need for transfusions, and possibly decrease the propensity of life threatening thrombosis. Eculizumab (h5G1.1-mAb) is a humanized monoclonal antibody that like CD59 inhibits terminal complement.

This study is an open label, multi-center study of eculizumab, administered intravenously for 52 weeks to approximately 85 PNH patients. The study is designed to evaluate the safety of eculizumab in transfusion dependent patients with paroxysmal nocturnal hemoglobinuria (PNH) and to determine if the administration of this terminal complement inhibitor could provide a safe and effective substitute for CD59 function.

ELIGIBILITY:
* INCLUSION CRITERIA
* The study population will comprise individuals who have transfusion-dependent hemolytic PNH.
* Each patient must meet the following criteria to be enrolled in this study:

  1. Individuals at least 18 years of age
  2. Patients with a diagnosis of PNH greater than 6 months
  3. Presence of a GPI deficient red blood cell clone (type III cells) by flow cytometry of greater than or equal to 10%
  4. Patients must have: at least one transfusion in the past two years for anemia or anemia-related symptoms -or personal beliefs that preclude the use of transfusion, with severe hemolytic PNH
  5. Documented LDH level greater than or equal to 1.5 x upper limit of normal (ULN) within 12 weeks of Visit 1 or during the Screening Period
  6. Patient must be willing and able to give written informed consent.
  7. Patients must avoid conception during the trial using a method that is most appropriate for their physical state and culture.
* Subjects must have a Visa allowing stay in United States for the duration of the study (up to 3 years).
* Subjects must provide documentation of residence during stay in the United States.
* The subject must be willing to keep all visits and not travel outside of the country while being treated under the protocol.
* The subject must understand that the drug may not be made commercially available in their country.
* Once the protocol and extension study is complete, the subject must come off study medication and it will not be made available to them if they return to their country.

EXCLUSION CRITERIA

-Any patient meeting any of the following criteria will be excluded from the study:

1. Platelet count of less than 30,000/mm3
2. Absolute Neutrophil count less than or equal to 500/uL
3. Presence or suspicion of active bacterial infection, in the opinion of the Investigator, at Visit 2 or recurrent bacterial infections
4. Known or suspected hereditary complement deficiency
5. History of bone marrow transplantation
6. Participation in any other investigational drug trial or exposure to other investigational agent, device, or procedure within 30 days prior to screening
7. Pregnant, breast-feeding, or intending to conceive during the course of the study,including the Safety Follow-up Visits

8 .History of meningococcal disease

9. Patients who are not vaccinated against N. meningitidis at least 14 days prior to Visit 2

10. Any condition that, in the opinion of the Investigator, could increase the patient's risk by participating in the study or confound the outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87
Dates: Start 2005-08-09; Study Completion 2007-06-25

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Walport MJ. Complement. First of two parts. N Engl J Med. 2001 Apr 5;344(14):1058-66. doi: 10.1056/NEJM200104053441406. No abstract available. PMID 11287977
- [Derived] Brodsky RA, Young NS, Antonioli E, Risitano AM, Schrezenmeier H, Schubert J, Gaya A, Coyle L, de Castro C, Fu CL, Maciejewski JP, Bessler M, Kroon HA, Rother RP, Hillmen P. Multicenter phase 3 study of the complement inhibitor eculizumab for the treatment of patients with paroxysmal nocturnal hemoglobinuria. Blood. 2008 Feb 15;111(4):1840-7. doi: 10.1182/blood-2007-06-094136. Epub 2007 Nov 30. PMID 18055865